CLINICAL TRIAL: NCT04951518
Title: VAN - Training of Emergency Medical Services to Improve Stroke Outcomes in Northwest Arkansas
Brief Title: VAN Assessment Tool in the Treatment of Acute Ischemic Stroke
Status: Completed | Type: Observational
Sponsor: Washington Regional Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: V-109
Record Dates: First submitted 2021-06-28; First posted 2021-07-06 (Actual); Last update posted 2022-04-27 (Actual); Status verified 2022-04

CONDITIONS: Acute Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 5 Days
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Van Positive: Large Vessel Occlusion Positive
  Interventions: Other: VAN Stroke Scale
- Van Negative: Large Vessel Occlusion Negative
  Interventions: Other: VAN Stroke Scale

INTERVENTIONS:
Other: VAN Stroke Scale — V.A.N Stroke Assessment measures unilateral weakness with visual deficits, aphasia, and neglect in possible stroke patients

SUMMARY:
To investigate the reliability of VAN tool as administered by Emergency Medical Services personnel to predict presence of a large vessel occlusion in setting of cerebral ischemic infarction

DETAILED DESCRIPTION:
The investigators propose to perform a 6-month pilot study in Northwest Arkansas in collaboration of two EMS providers; Central EMS and AirEvac. These local providers operate in the WRMC catchment area and transport over 90% of patients with a suspected stroke to WRMC comprehensive stroke center. Thus no changes to their standard operations would be implemented. The aim of this pilot study would be to test the accuracy of VAN-screening in the area in patients treated at WRMC - thus only patients who are brought to WRMC as per current protocol would be included in the study.

The investigators would train Central EMS and AirEvac personnel to perform the V.A.N screen, over a 2-month period (estimated June-July 2020) in several sessions at the Central EMS training center at 800 S. School Ave. in Fayetteville. This training would be performed by study investigators, assisted by medical students, residents, and advanced practice nurses (APNs). The training would consist of a training video, hands-on instruction, and sample scenarios.The investigators would survey all training participants to gather feedback on the format, delivery, and understanding of the training material. The PowerPoint presentation planned for the training session, as well as the post-training quiz, are attached as Appendices to this application. The investigators would expect a rate of 80% correct answers in the post-training quiz. All questions and scenarios would be discussed with all trainees after the quiz, and re-takes would be allowed.

ELIGIBILITY:
Inclusion Criteria:

* Patients treated for stroke at WRMC who are transported to the hospital by Central EMS or AirEvac

Exclusion Criteria:

* Stroke patients who arrive directly to the hospital (without the use of EMS services)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Anyone experiencing acute ischemic stroke symptoms
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2020-10-22 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-03-17 (Actual)

PRIMARY OUTCOMES:
Reliability of VAN Assessment Tool | 1 Year
  To investigate the reliability of VAN tool as administered by Emergency Medical Services personnel to predict presence of a large vessel occlusion in setting of cerebral ischemic infarction

SECONDARY OUTCOMES:
Eligibility for Thrombolysis | 1 Year
  To investigate effect of the VAN tool to predict persons eligible for thrombolysis
Eligibility for Thrombectomy | 1 Year
  To investigate effect of the VAN tool to predict persons eligible for thrombectomy
Door to Intervention Time | 1 Year
  To investigate the effect of prehospital notification of VAN positive status vs routine notification on time door to needle or door to thrombectomy time
Modified Rankin Score | 1 Year
  To compare the discharge disposition and Rankin score of patients post intervention with VAN prenotification vs routine notification. Rankin scores ranging from 0 - 5, with 0 being fully functioning and independent, and 5 being severe disability requiring constant nursing care.

CONTACTS AND LOCATIONS:
Locations (1):
- Washington Regional Medical Center, Fayetteville, Arkansas, United States

IPD SHARING:
Plan to Share IPD: No